CLINICAL TRIAL: NCT00721175
Title: Efficacy and Cost Analysis of Plastic Stent Compare to Metallic Stent in Unresectable Complex Hilar Cholangiocarcinoma; a Randomized Controlled Trial
Brief Title: Efficacy and Cost Analysis of Plastic Stent Compare to Metallic Stent in Hilar Cholangiocarcinoma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Apichat Sangchan, Assist. Prof., Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HE500636
Record Dates: First submitted 2008-07-21; First posted 2008-07-23 (Estimated); Results first posted 2011-12-23 (Estimated); Last update posted 2011-12-23 (Estimated); Status verified 2011-11

CONDITIONS: Hilar Cholangiocarcinoma
Keywords: biliary stent; plastic stent; metallic stent; Complex hilar cholangiocarcinoma (Bismuth type II,III,IV)
MeSH Terms: conditions — Klatskin Tumor | interventions — Self Expandable Metallic Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SEMS (Experimental): self-expandable metal stent group
  Interventions: Device: biliary stent (self expandable metallic stent)
- PS (Active Comparator): plastic stent group
  Interventions: Device: PS

INTERVENTIONS:
Device: biliary stent (self expandable metallic stent) — metallic stent was inserted into right or left hepatic duct which was planed before intervention using CT scan or MRCP
  Other Names: self expandable metallic stent
  Arms: SEMS
Device: PS — plastic stent was inserted into right or left hepatic duct which was planed before intervention using CT scan or MRCP
  Other Names: Amsterdam type plastic stent
  Arms: PS

SUMMARY:
The purpose of this study is to compare the adequacy of unilateral endoscopic biliary drainage using metallic stent with plastic stent in unresectable, complex, hilar, cholangiocarcinoma and cost analysis.

DETAILED DESCRIPTION:
There are two types of biliary stents: 1) the plastic stent made from polyethylene or polytetrafluoroethylene; and, 2) the metal stent braided in the form of a tubular mesh from surgical-grade stainless steel alloy and designed to expand to a maximum diameter of 10 mm. The main drawback of the plastic stent is the relatively high occlusion rate, but its advantage is the lower cost. The use of a metal stent for hilar tumor has many theoretical advantages: 1) the flexible open-mesh design should allow drainage of secondary duct branches; and, 2) its larger diameter may provide better drainage and longer patency (~3-9 months).

Whether one type of stent is superior in terms of adequacy of drainage or cost-effectiveness remains undefined. Therefore, we would conduct this study to assess the efficacy of drainage of endoscopically-inserted, unilateral, plastic stents vs. metallic stents in unresectable, complex, hilar cholangiocarcinoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable complex hilar cholangiocarcinoma which diagnosis and staging based on computed tomography(CT) or magnetic resonance cholangiopancreatography (MRCP)

Exclusion Criteria:

* Patients with ASA 4 or 5
* Patients with liver failure.
* Patients unable to comply with follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2007-11; Primary Completion 2010-04 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: apichat sangchan, MD, Principal Investigator — Department of Medicine. Faculty of Medicine. KhonKaen University
Locations (1):
- Srinagarind Hospital. KhonKaen University., Muang, KhonKaen, Thailand

REFERENCES:
- [Background] De Palma GD, Pezzullo A, Rega M, Persico M, Patrone F, Mastantuono L, Persico G. Unilateral placement of metallic stents for malignant hilar obstruction: a prospective study. Gastrointest Endosc. 2003 Jul;58(1):50-3. doi: 10.1067/mge.2003.310. PMID 12838220
- [Background] Wagner HJ, Knyrim K, Vakil N, Klose KJ. Plastic endoprostheses versus metal stents in the palliative treatment of malignant hilar biliary obstruction. A prospective and randomized trial. Endoscopy. 1993 Mar;25(3):213-8. doi: 10.1055/s-2007-1010295. PMID 7686100
- [Background] Freeman ML, Overby C. Selective MRCP and CT-targeted drainage of malignant hilar biliary obstruction with self-expanding metallic stents. Gastrointest Endosc. 2003 Jul;58(1):41-9. doi: 10.1067/mge.2003.292. PMID 12838219
- [Derived] Sangchan A, Kongkasame W, Pugkhem A, Jenwitheesuk K, Mairiang P. Efficacy of metal and plastic stents in unresectable complex hilar cholangiocarcinoma: a randomized controlled trial. Gastrointest Endosc. 2012 Jul;76(1):93-9. doi: 10.1016/j.gie.2012.02.048. Epub 2012 May 15. PMID 22595446
- See also: KhonKaen University Ethics Committee for Human Research — http://eckku.kku.ac.th/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between November 2007 and March 2010, one hundred and eight patients who visited medical clinic at Srinagarind hospital, Khon Kaen University were randomized into the study
Pre-assignment Details: the patients were excluded from trial after enrollment if CBD canulation is failed.
Groups:
- Plastic Stent: plastic stent group
Period: Overall Study
Arm/Group | SEMS | Plastic Stent
Started | 54 | 54
Completed | 54 | 54
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SEMS | Plastic Stent | Total
Number analyzed (Participants) | 54 | 54 | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49 | 49 | 98
  >=65 years | 5 | 5 | 10
Age Continuous [Mean (Standard Deviation); unit: years] | 62.7 (10.3) | 57.3 (11.7) | 60.0 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 43 | 43 | 86
Region of Enrollment [Number; unit: participants]
  Thailand | 54 | 54 | 108

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Adequate Biliary Drainage in Metallic Stent and Plastic Stent Group.(ITT Analysis)
Description: Successful drainage was defined as a decrease in total bilirubin level to less than 30% or 50% of pretreatment level within two and four weeks respectively in each patient.
Time Frame: at 2 weeks and 4 weeks after stent insertion
Population: All 108 participants enrolled into the study were analyzed based on ITT analysis basis.(54 participants in each group)
Measure: Mean (95% Confidence Interval); unit: proportion of participants
Groups:
- SEMS: SEMS (Self-expandable metal stent group)
Arm/Group | SEMS | Plastic Stent
Number analyzed (Participants) | 54 | 54
proportion of participants | .7037037 [.5819144 to .825493] | .46296 [.3299707 to .5959553]
Statistical Analysis 1: Comparison: SEMS vs Plastic Stent; Test type: Superiority or Other; p = 0.011, Two-sample test of proportion; Mean Difference (Final Values) = -.2407407, 95% CI 2-sided [-.4210726 to -.0604089], Standard Error of Mean .0920078

2. Secondary Outcome: Patients Survival Times
Description: survival times of the patients after the first stent insertion
Time Frame: until patient died or 6 months after the last patient was enrolled
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | SEMS | Plastic Stent
Number analyzed (Participants) | 54 | 54
days | 126 [42 to 290] | 49 [21 to 97]
Statistical Analysis 1: Comparison: SEMS vs Plastic Stent; Test type: Superiority or Other; p = 0.0021, Log Rank

3. Secondary Outcome: Cost Effective Ratio of Metallic and Plastic Stent
Description: cost per quality adjusted life year (QALY)of metallic stent and plastic stent calculated from Markov model using transitional probabilities, cost and utilities from this study and the available literature
Time Frame: until the patients expire (Markov model)
Population: Simulation cohort of any number of the patients (1, 100 or 1,000 patients) enter the Markov model using transitional probabilities, cost data, utility data from this study and available literature to calculate the cost effectiveness ratio of metallic stent and plastic stent in unresectable complex hilar cholangiocarcinoma
Measure: Number; unit: cost (US$) per QALY
Arm/Group | SEMS | Plastic Stent
Number analyzed (Participants) | 1 | 1
cost (US$) per QALY | 10742 | 19085

4. Primary Outcome: Proportion of Patients With Adequate Biliary Drainage in Metallic Stent and Plastic Stent Group.(Per Protocol Analysis)
Description: Successful drainage was defined as a decrease in total bilirubin level to less than 30% or 50% of pretreatment level within two and four weeks respectively.
Time Frame: at 2 weeks and 4 weeks after stent insertion
Population: 91 participants who had successful stent insertion were analyzed based on per protocol analysis.
Measure: Mean (95% Confidence Interval); unit: proportion of participants
Arm/Group | SEMS | Plastic Stent
Number analyzed (Participants) | 45 | 46
proportion of participants | 0.822 [0.711 to 0.934] | 0.543 [0.400 to 0.687]
Statistical Analysis 1: Comparison: SEMS vs Plastic Stent; Test type: Superiority or Other; p = 0.004, Two-sample test of proportion; Mean Difference (Final Values) = -.278744, 95% CI 2-sided [-.4609466 to -.0965414], Standard Error of Mean .0929622

ADVERSE EVENTS:
Arm/Group | SEMS | Plastic Stent
Serious Adverse Events (participants affected / at risk) | 14/54 | 21/54
Other Adverse Events (participants affected / at risk) | 0/54 | 1/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SEMS (N=54) | Plastic Stent (N=54)
cholangitis (Hepatobiliary disorders) | 8 (8) | 13 (13)
pancreatitis (Hepatobiliary disorders) | 8 | 8
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SEMS (N=54) | Plastic Stent (N=54)
sphicterotomy bleeding (Hepatobiliary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No